CLINICAL TRIAL: NCT01996241
Title: Evaluation of an Intervention Supporting Adolescent Girls From Marginalized Communities to Complete Secondary Schooling
Brief Title: Evaluation of an Intervention for Adolescent Girls in Karnataka
Acronym: Samata
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karnataka Health Promotion Trust (Other)
Collaborators: University of Manitoba (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 111/2013
Record Dates: First submitted 2013-11-16; First posted 2013-11-27 (Estimated); Results first posted 2019-09-25 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Secondary School Entry and Completion; Child Marriage
Keywords: adolescent girls; female sex work; age at marriage; retention in school; sexual debut; India; Karnataka

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Village Clusters (Experimental): Receive multi-level, structural and norms-based intervention
  Interventions: Behavioral: Multi-level, structural and norms-based intervention
- Control Village Clusters (No Intervention): No multi-level, structural and norms-based intervention

INTERVENTIONS:
Behavioral: Multi-level, structural and norms-based intervention — Receive multi-level, structural and norms-based intervention
  Arms: Intervention Village Clusters

SUMMARY:
This cluster Randomised Control Trial is evaluating an intervention to support adolescent girls from marginalised communities in northern Karnataka State, South India to complete secondary school, thereby reducing their vulnerability to HIV infection from early marriage and entry into sex work at young ages. The intervention will test innovations to address both supply and demand side barriers to girls' completion of secondary school, and will have long-term educational and livelihood benefits, in addition to reducing vulnerability to HIV.

School-based constraints will be addressed by improving academic outcomes through teacher training and academic support to students; addressing gender-related and skill-based gaps among teachers; training of local female teachers; and increasing the content knowledge of secondary school teachers. Demand side barriers will be addressed by reducing economic pressures that households face to withdraw girls' from school; building appreciation and value of girls' education; building family and community accountability for school attendance; creating safe spaces for girls and strengthening their agency; and engaging boys in promoting and supporting girls' education.

Primary stakeholders will include teachers and students, especially adolescent girls in the school (7th to 10 the standard) from marginalized communities. Secondary stakeholders will include school development and management committees (SDMCs), families, boys and the communities that are served by the schools. 80 village clusters (40 intervention; 40 control) were randomly selected from 125 village clusters in Bagalkote and Vijayapura districts. The intervention will be implemented with village communities and high schools in 40 village clusters in Bagalkote and Vijayapura districts. The intervention will be implemented in collaboration with the Department of State Educational Research and Training (DSERT), Karnataka; the Adolescent Education Cell, Government College of Teachers' Education (CTE), Jamkhandi; and the Institute for Advanced Studies in Education (IASE), Gulbarga.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent girls in Standard 7

Exclusion Criteria:

* None

Ages: 13 Years to 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2457 (Actual)
Dates: Start 2014-01; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shajy Isac, PhD, Study Director — Karnataka Health Promotion Trust
Locations (1):
- Bagalkot and Bijapur Districts, Bagalkot, Karnataka, India

IPD SHARING:
Plan to Share IPD: Yes
Data will be anonymised and made available for secondary analyses on request, following publication of trial findings.

REFERENCES:
- [Background] Beattie TS, Bhattacharjee P, Isac S, Davey C, Javalkar P, Nair S, Thalinja R, Sudhakar G, Collumbien M, Blanchard JF, Watts C, Moses S, Heise L. Supporting adolescent girls to stay in school, reduce child marriage and reduce entry into sex work as HIV risk prevention in north Karnataka, India: protocol for a cluster randomised controlled trial. BMC Public Health. 2015 Mar 25;15:292. doi: 10.1186/s12889-015-1623-7. PMID 25881037
- [Background] Ramanaik S, Collumbien M, Prakash R, Howard-Merrill L, Thalinja R, Javalkar P, Murthy S, Cislaghi B, Beattie T, Isac S, Moses S, Heise L, Bhattacharjee P. Education, poverty and "purity" in the context of adolescent girls' secondary school retention and dropout: A qualitative study from Karnataka, southern India. PLoS One. 2018 Sep 5;13(9):e0202470. doi: 10.1371/journal.pone.0202470. eCollection 2018. PMID 30183747
- [Background] Mazzuca A, Nagarchi D, Ramanaik S, Raghavendra T, Javalkar P, Rotti S, Bhattacharjee P, Isac S, Cohen A, Beattie T. Developing a Mental Health Measurement Strategy to Capture Psychological Problems among Lower Caste Adolescent Girls in Rural, South India. Transcult Psychiatry. 2019 Feb;56(1):24-47. doi: 10.1177/1363461518789540. Epub 2018 Aug 16. PMID 30113275
- [Background] Prakash R, Beattie T, Javalkar P, Bhattacharjee P, Ramanaik S, Thalinja R, Murthy S, Davey C, Blanchard J, Watts C, Collumbien M, Moses S, Heise L, Isac S. Correlates of school dropout and absenteeism among adolescent girls from marginalized community in north Karnataka, south India. J Adolesc. 2017 Dec;61:64-76. doi: 10.1016/j.adolescence.2017.09.007. Epub 2017 Sep 29. PMID 28968543
- [Background] Bhagavatheeswaran L, Nair S, Stone H, Isac S, Hiremath T, Thalinda R, Vadde K, Doddamane M, Srikantamurthy HS, Heise L, Watts C, Schweisfurth M, Bhattacharjee P, Beattie TS. The barriers and enablers to education among scheduled caste and scheduled tribe adolescent girls in northern Karnataka, South India: A qualitative study. Int J Edu Dev. 2016. 49 262-270
- [Derived] Prakash R, Beattie TS, Cislaghi B, Bhattacharjee P, Javalkar P, Ramanaik S, Thalinja R, Davey C, Gafos M, Watts C, Collumbien M, Moses S, Isac S, Heise L. Changes in Family-Level Attitudes and Norms and Association with Secondary School Completion and Child Marriage Among Adolescent Girls: Results from an Exploratory Study Nested Within a Cluster-Randomised Controlled Trial in India. Prev Sci. 2020 Nov;21(8):1065-1080. doi: 10.1007/s11121-020-01143-1. PMID 32720188
- [Derived] Prakash R, Beattie TS, Javalkar P, Bhattacharjee P, Ramanaik S, Thalinja R, Murthy S, Davey C, Gafos M, Blanchard J, Watts C, Collumbien M, Moses S, Heise L, Isac S. The Samata intervention to increase secondary school completion and reduce child marriage among adolescent girls: results from a cluster-randomised control trial in India. J Glob Health. 2019 Jun;9(1):010430. doi: 10.7189/jogh.09.010430. PMID 31448111
- [Derived] Beattie TS, Prakash R, Mazzuca A, Kelly L, Javalkar P, Raghavendra T, Ramanaik S, Collumbien M, Moses S, Heise L, Isac S, Watts C. Prevalence and correlates of psychological distress among 13-14 year old adolescent girls in North Karnataka, South India: a cross-sectional study. BMC Public Health. 2019 Jan 10;19(1):48. doi: 10.1186/s12889-018-6355-z. PMID 30630455
- See also: Link to Samata Trial Protocol Paper — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4391662/pdf/12889_2015_Article_1623.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 80 of 121 village clusters in Vijayapura and Bagalkote districts, Karnataka State, were randomly selected (40 intervention; 40 control). Girls were recruited from two successive academic years (cohorts 1 and 2) to increase study power and achieve required sample size. Analysis was planned by trial arm rather than separately for two study cohorts.
Units Other Than Participants: Village cluster
Groups:
- Intervention Village Cluster: All SC/ST girls in final year of primary school living in intervention villages eligible for study enrolment.
- Control Village Cluster: All SC/ST girls in final year of primary school living in control villages eligible for study enrolment
Period: Overall Study
Arm/Group | Intervention Village Cluster | Control Village Cluster
Started | 1164; 40 Village cluster | 1111; 40 Village cluster
Completed | 912; 40 Village cluster | 876; 40 Village cluster
Not Completed | 252; 0 Village cluster | 235; 0 Village cluster
Not completed — Lost to Follow-up | 252 | 235

BASELINE CHARACTERISTICS:
Population: Of the total population of SC/ST girls in the final year of primary school who were eligible for this study, 1164/1265 in the intervention arm and 1111/1192 in the control arm participated in the baseline survey. 101 girls from the intervention and 81 from the control were not surveyed at baseline.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Village Cluster | Control Village Cluster | Total
Number analyzed (Participants) | 1164 | 1111 | 2275
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 13.0 [12 to 16] | 13.0 [12 to 15] | 13.0 [12 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1164 | 1111 | 2275
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  India | 1164 | 1111 | 2275
District [Count of Participants; unit: Participants]
  Bagalkote | 639 | 620 | 1259
  Vijapura | 525 | 491 | 1016
Caste (ST vs. SC) [Count of Participants; unit: Participants]
  Scheduled Tribe | 278 | 209 | 487
  Schedued Caste | 886 | 902 | 1788
Non-literate Household Head [Count of Participants; unit: Participants] | 748 | 667 | 1415
Village Type (Feeder vs. Main) [Count of Participants; unit: Participants]
  Feeder Village | 321 | 346 | 667
  Main Village | 843 | 765 | 1608
Household wealth quintile (Poorest) [Count of Participants; unit: Participants] | 228 | 227 | 455
Devadasi Family [Count of Participants; unit: Participants] | 65 | 47 | 112

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Completing Secondary School [Sit 10th Standard Exam]
Description: This outcome will be assessed using data collected from all study participants at end-line, using the face-to-face questionnaire.
Time Frame: May-August 2016 (cohort one) and May-August 2017 (cohort two)
Measure: Count of Participants; unit: Participants
Groups:
- SC/ST Girls in Intervention Village Cluster: All SC/ST girls in final year of primary school living in intervention villages eligible for study enrolment.
- SC/ST Girls in Control Village Cluster: All SC/ST girls in final year of primary school living in control villages eligible for study enrolment
Arm/Group | SC/ST Girls in Intervention Village Cluster | SC/ST Girls in Control Village Cluster
Number analyzed (Participants) | 912 | 876
Participants | 680 | 658
Statistical Analysis 1: Comparison: SC/ST Girls in Intervention Village Cluster vs SC/ST Girls in Control Village Cluster; Test type: Other — Odds ratio (95% CI), p-value for all the outcomes; p = 0.98, Regression, Logistic — Adjusted models controlled for cluster, village strata, village type, caste, household literacy status, stratum (individual-level data endline) and poor learning environment at school, school dropout, and marriage (cluster-level summaries baseline); Mixed-effects; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.7 to 1.38]

2. Primary Outcome: Number of Participants Married [by Trial End Line]
Description: as for outcome 1
Time Frame: May-August 2016 (cohort one) and May-August 2017 (cohort two)
Measure: Count of Participants; unit: Participants
Arm/Group | SC/ST Girls in Intervention Village Cluster | SC/ST Girls in Control Village Cluster
Number analyzed (Participants) | 912 | 876
Participants | 92 | 84
Statistical Analysis 1: Comparison: SC/ST Girls in Intervention Village Cluster vs SC/ST Girls in Control Village Cluster; Test type: Other; p = 0.98, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Mixed-effects; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.7 to 1.4]

3. Secondary Outcome: Number of Participants Entering Into 8th Standard [Start Secondary School]
Description: Due to delays at the start of the cluster-Randomized Controlled Trial, the intervention had not started when cohort one girls were interviewed. This outcome will be assessed using data from cohort two girls only, using the face-to-face questionnaire. To reduce recall bias, we will use data collected at the first interview (baseline) to measure this outcome.
Time Frame: March-May 2014
Population: outcome assessed using data from cohort two girls only, using the baseline face-to-face questionnaire.
Measure: Count of Participants; unit: Participants
Groups:
- SC/ST Girls in Intervention Village Cluster: All SC/ST girls in cohort 2 in final year of primary school living in intervention villages
- SC/ST Girls in Control Village Cluster: All SC/ST girls in cohort 2 in final year of primary school living in control villages
Arm/Group | SC/ST Girls in Intervention Village Cluster | SC/ST Girls in Control Village Cluster
Number analyzed (Participants) | 625 | 566
Participants | 580 | 516
Statistical Analysis 1: Comparison: SC/ST Girls in Intervention Village Cluster vs SC/ST Girls in Control Village Cluster; Test type: Other; p = 0.331, Regression, Logistic — Adjusted for village strata and cluster, village type, caste, household literacy status, stratum using individual-level data and poor learning environment at school, school dropout, and marriage (in the form of cluster-level summaries); Mixed-effects; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.2 to 2.31]

4. Secondary Outcome: Number of Participants Passing 10th Standard [Pass 10th Standard Exam]
Description: as for outcome 1
Time Frame: May-August 2016 (cohort one) and May-August 2017 (cohort two)
Measure: Count of Participants; unit: Participants
Arm/Group | SC/ST Girls in Intervention Village Cluster | SC/ST Girls in Control Village Cluster
Number analyzed (Participants) | 912 | 876
Participants | 518 | 530
Statistical Analysis 1: Comparison: SC/ST Girls in Intervention Village Cluster vs SC/ST Girls in Control Village Cluster; Test type: Other; p = 0.26, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Mixed-effects; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.6 to 1.15]

5. Secondary Outcome: Number of Participants Having Sexual Debut [by Trial End Line]
Description: This outcome will be assessed using data collected from all study participants at end-line, using the self-completed questionnaire.
Time Frame: May-August 2016 (cohort one) and May-August 2017 (cohort two)
Measure: Count of Participants; unit: Participants
Arm/Group | SC/ST Girls in Intervention Village Cluster | SC/ST Girls in Control Village Cluster
Number analyzed (Participants) | 912 | 876
Participants | 64 | 53
Statistical Analysis 1: Comparison: SC/ST Girls in Intervention Village Cluster vs SC/ST Girls in Control Village Cluster; Test type: Other; p = 0.79, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Mixed-effects; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.7 to 1.55]

6. Secondary Outcome: Number of Participants Married and Co-habiting With Husband [by Trial End Line]
Description: as for outcome 1
Time Frame: May-August 2016 (cohort one) and May-August 2017 (cohort two)
Measure: Count of Participants; unit: Participants
Arm/Group | SC/ST Girls in Intervention Village Cluster | SC/ST Girls in Control Village Cluster
Number analyzed (Participants) | 912 | 876
Participants | 43 | 46
Statistical Analysis 1: Comparison: SC/ST Girls in Intervention Village Cluster vs SC/ST Girls in Control Village Cluster; Test type: Other; p = 0.45, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Mixed-effects; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.5 to 1.34]

ADVERSE EVENTS:
Time Frame: 3 years, 6 months
Arm/Group | SC/ST Girls in Intervention Village Cluster | SC/ST Girls in Control Village Cluster
All-Cause Mortality (participants affected / at risk) | 0/1265 | 0/1192
Serious Adverse Events (participants affected / at risk) | 0/1265 | 0/1192
Other Adverse Events (participants affected / at risk) | 0/1265 | 0/1192

LIMITATIONS AND CAVEATS:
Due to funding delays at the start of the trial, the intervention started later than planned, when girls in cohort 1 were in second year of secondary school and girls in cohort 2 were in first term of secondary school.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT01996241/SAP_000.pdf
  • Study Protocol (2014-11-18): https://cdn.clinicaltrials.gov/large-docs/41/NCT01996241/Prot_001.pdf